CLINICAL TRIAL: NCT00005611
Title: Phase I Study of BMS-188797 in Patients With Advanced Malignancies
Brief Title: BMS-188797 in Treating Patients With Advanced Solid Tumors That Have Not Responded to Previous Treatment
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067740; MCC-11836; BMS-CA159-001; MCC-IRB-5140; NCI-G00-1744
Record Dates: First submitted 2000-05-02; First posted 2004-07-26 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2000-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — BMS188797

INTERVENTIONS:
Drug: BMS-188797

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of BMS-188797 in treating patients who have advanced solid tumors that have not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and recommended phase II dose, dose limiting toxicities, and safety of BMS-188787 in patients with nonhematologic malignancies. II. Determine the plasma pharmacokinetics of BMS-188797 in these patients. III. Describe any antitumor activity of this treatment in these patients.

OUTLINE: This is a dose escalation study. Patients receive BMS-188797 IV over 1 hour. Treatment continues every 21 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of BMS-188797 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities. Patients are followed every 4 weeks until toxicities resolve, and then at the investigator's discretion.

PROJECTED ACCRUAL: Approximately 20-40 patients will be accrued for this study over 12-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed nonhematologic malignancy unresponsive to existing therapy or for which no curative therapy exists Patients with prostate cancer must have withdrawn from antiandrogen therapy (flutamide, bicalutamide) for at least 4 weeks and must have progressive disease Measurable or evaluable disease No active brain metastases (e.g., cerebral edema, progression from prior imaging study, requirement for steroids, or clinical symptoms)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL ALT and AST no greater than 2.5 times upper limit of normal (ULN) (unless due to hepatic metastases) Renal: Creatinine less than 1.5 times ULN Other: No serious uncontrolled medical disorder or active infection that would preclude study No hypersensitivity to agents containing polyoxyethylated castor oil (Cremophor EL) except in patients who received prior taxane therapy with premedication and did not experience greater than grade 1 hypersensitivity reaction Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since prior nitrosoureas, mitomycin, or carboplatin) Prior taxanes allowed No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 2 weeks since prior hormonal therapy No concurrent steroids No concurrent hormonal therapy (except leuprolide acetate for prostate cancer) Radiotherapy: At least 4 weeks since prior radiotherapy to 30% or more of bone marrow No concurrent radiotherapy Surgery: Not specified Other: No other concurrent investigational anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: William S. Dalton, MD, PhD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute